CLINICAL TRIAL: NCT04457700
Title: Computed Tomography-based Radiomics of Axillary Lymph Node Pathological Complete Remission (ypN0) in Breast Cancer Undergoing Neoadjuvant Chemotherapy
Brief Title: CT-based Radiomics of ALN pCR (ypN0) in Breast Cancer Undergoing NAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Tao OUYANG, Director of Breast Center of Peking University Cancer Hospital, Peking University
Other Study IDs: BCP28
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Triple-negative Breast Cancer; HER2-positive Breast Cancer
Keywords: Breast cancer; Neoadjuvant chemotherapy; Lymph node; Radiomic; Pathologic complete remission
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms; Pathologic Complete Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Axillary lymph node status are determined in FNA/CNB and surgical specimen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Triple-negative and HER2 Positive breast cancer: Patients with triple-negative or HER2 Positive breast cancer, axillary lymph node metastasis who underwent NAC are eligible for this study. Axillary lymph node metastasis is confirmed by fine needle aspiration (FNA) or core needle biopsy (CNB) at initial diagnosis. CT-based radiomics will be uesd in evaluating the response and predicting pCR of metastatic lymph nodes after NAC in breast cancer patients.

SUMMARY:
This is a prospective, single-center, non-randomized, non-controlled observational study.

DETAILED DESCRIPTION:
Almost 55-62% of patients with triple-negative or human epidermal growth factor receptor 2 (HER2) positive, node-positive breast cancer achieve an axillary pathologic complete remission (pCR) after neoadjuvant chemotherapy (NAC). To avoid surgery post-NAC, it is paramount to accurately identify patients who achieve pCR in axillary lymph node (ALN). We found that patients with normal-appearing lymph nodes on computed tomography (CT) based radiomics of the axilla after chemotherapy had a lower risk of developing residual nodal disease. However, the features of CT-based radiomics for pCR ALN following NAC has not been established yet. This study aimed to assess the performance of CT-based radiomics in evaluating the response and predicting pCR of metastatic lymph nodes after NAC in breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Triple-negative or HER2-positve invasive breast cancer with axillary lymph node metastasis by confirmed by fine needle aspiration or core needle biopsy.
* Underwent computed tomography for assessment of axillary lymph node status before and after neoadjuvant chemotherapy.
* Attend the study voluntarily, sign the informed consent.

Exclusion Criteria:

* Contradiction for adjuvant chemotherapy.
* Contradiction for proceeding surgery.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Triple-negative or HER2-positve invasive breast cancer with axillary lymph node metastasis: stage T1-3N1-2M0.
Sampling Method: Probability Sample
Enrollment: 218 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
The features of CT-based radiomics for axillary lymph node achieved pCR after neoadjuvant chemotherapy | within 8 weeks after obtaining the post-surgery pathological results
  Sensitivity, specificity, positive-predictive value (PPV) and negative-predictive value (NPV) of CT-based radiomics for axillary lymph node status after neoadjuvant chemotherapy will be assessed.

SECONDARY OUTCOMES:
Receiver operating characteristic (ROC) curve analysis | within 8 weeks after obtaining the post-surgery pathological results
  The diagnostic performance of CT-based radiomics for the evaluation of ALN after NAC was evaluated with receiver operating characteristic (ROC) curve analysis. The diagnostic accuracy was estimated by calculating the area under the ROC curve

CONTACTS AND LOCATIONS:
Overall Officials: Lize Wang, MD, Principal Investigator — Breast center at Peking University Cancer Hospital
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided